CLINICAL TRIAL: NCT06897150
Title: Efficacy and Safety of Carotegrast Methyl in Active Ulcerative Colitis: A Real-World Prospective Cohort Study
Brief Title: Carotegrast Methyl in Ulcerative Colitis
Acronym: CAR in UC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Takayuki Yamamoto (Other)
Responsible Party: Sponsor-Investigator, Takayuki Yamamoto, The Director of the Hospital, Yokkaichi Hazu Medical Center
Organization: Yokkaichi Hazu Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Yokkaichi Hazu 2024-11
Record Dates: First submitted 2025-03-19; First posted 2025-03-26 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — AJM300

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Carotegrast methyl (Experimental): Carotegrast methyl at a dosage of 960 mg three times daily
  Interventions: Drug: Carotegrast methyl

INTERVENTIONS:
Drug: Carotegrast methyl — a dosage of 960 mg three times daily

SUMMARY:
Carotegrast methyl, an oral α4-integrin inhibitor, was recently approved in Japan for the treatment of active ulcerative colitis (UC). However, real-world data regarding its efficacy and safety remain scarce. This study aimed to assess the clinical effectiveness and safety profile of carotegrast methyl in patients with active UC.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with UC based on endoscopic and histological findings
* Patients with clinically and endoscopically moderate UC who were eligible for outpatient treatment (however, patients in clinical remission or with mild clinical activity but endoscopically moderate UC were also considered eligible as an exception)
* Patients who exhibited an inadequate response to or intolerance of 5-ASA formulations (including topical agents) or budesonide formulations (including topical agents)
* Patients who provided informed consent for endoscopic examinations at the start of treatment and during the treatment period
* Patients who agreed to blood sampling and fecal biomarker tests

Exclusion Criteria:

* Patients with severe disease on endoscopy (presumed ineffective due to the drug's characteristics)
* Patients currently using biologics, JAK inhibitors, thiopurines, or calcineurin inhibitors (tacrolimus or cyclosporine)
* Patients with a history of malignancy
* Patients with severe hepatic dysfunction
* Pregnant women or those planning pregnancy
* Patients with acute severe conditions, such as toxic megacolon, sepsis, peritonitis, or infectious colitis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 50 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2025-03-15 (Actual); Study Completion 2025-03-15 (Actual)

PRIMARY OUTCOMES:
Clinical remission | Week 8
  A total clinical subscores in the Mayo score of 0

SECONDARY OUTCOMES:
Endoscopic remission | Week 8
  Endoscopic subscore in the Mayo score of 0

OTHER OUTCOMES:
Clinical improvement | Week 24
  Decreae of clinical score in the mayo score at least 1

CONTACTS AND LOCATIONS:
Overall Officials: Takayuki Yamamoto, MD, PhD, Study Chair — Yokkaichi Hazu Medical Center; Takayuki Yamamoto, MD, PhD, Study Director — Yokkaichi Hazu Medical Center; Takayuki Yamamoto, MD, PhD, Principal Investigator — Yokkaichi Hazu Medical Center
Locations (1):
- Yokkaichi Hazu Medical Center, Yokkaichi, Mie-ken, Japan

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Within 6 months of the publication of study results Data will be available for access for 1 year
Access Criteria: The data will be available for use in further scientific research, such as additional analyses, validating clinical outcomes, or investigating new treatment options.
URL: https://yokkaichi.jcho.go.jp/